CLINICAL TRIAL: NCT00148564
Title: Energy Homeostasis and Metabolism in Patients With Schizophrenic Disorders Under Treatment With Atypical Antipsychotics
Brief Title: Energy Homeostasis Under Treatment With Atypical Antipsychotics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Martin Schaefer, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Energy
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2008-09-29 (Estimated); Status verified 2008-09

CONDITIONS: Schizophrenia
Keywords: weight gain; schizophrenia; atypical antipsychotics
MeSH Terms: conditions — Schizophrenia; Weight Gain | interventions — Olanzapine; ziprasidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olanzapine (Active Comparator)
  Interventions: Drug: olanzapine
- Zpirasidone (Active Comparator)
  Interventions: Drug: Ziprasidone

INTERVENTIONS:
Drug: olanzapine — treatment with either Olanzapine or Ziprasidone
  Other Names: Zyprexa
  Arms: Olanzapine
Drug: Ziprasidone — treatment with either Olanzapine or Ziprasidone
  Other Names: Zeldox
  Arms: Zpirasidone

SUMMARY:
The purpose of this study is to evaluate the effects of different atypical antipsychotics on weight changes, energy homeostasis, metabolism, energy intake as well as activity.

Patients with schizophrenia or schizoaffective disorders will be randomly assigned to be treated with ziprasidone or olanzapine for 24 weeks.

Primary outcome parameter are the weight changes after 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or related disorders(DSM-IV)
* Indication for long-term treatment with antipsychotics
* BMI between 20 to 30
* Weight changes less than 3kg in the last 3 months before inclusion
* Informed consent

Exclusion Criteria:

* Psychiatric comorbidity
* Depot antipsychotic in the last 2 months
* Antipsychotics in the last 2 weeks
* Treatment with olanzapine, clozapine or ziprasidone in teh last 3 months
* Treatment with drugs, that may lead to weight changes
* Significant endocrine, neurological, cardiovascular, hepatic, renal, metabolic, or other medical diseases or any clinically relevant abnormalities in laboratory tests
* Female subjects during pregnancy and breastfeeding
* Female subjects within childbearing years who were not using adequate birth control
* Patients who are judged by the investigator to be at serious suicide risk

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2004-03; Primary Completion 2007-03 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Primary outcome parameter are the weight changes after 24 weeks between olanzapine and ziprasidone treatment | during treatment

SECONDARY OUTCOMES:
Changes in energy homeostasis, food intake, metabolism | during and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schaefer, MD, Principal Investigator — Charite Campus Mitte; Dept. of Psychiatry and Psychotherapy and Department of Psychiatry, Kliniken Essen-Mitte
Locations (1):
- Charité Universitaetsmedizin Berlin; Campus Charité Mitte; Dept. for Psychiatry and Psychotherapy, Berlin, Germany